CLINICAL TRIAL: NCT04982471
Title: Connect® Lymphoma Disease Registry: A US-Based Prospective Observational Cohort Study
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NDS-DLBCL-003
Record Dates: First submitted 2021-07-20; First posted 2021-07-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular
Keywords: Non-Hodgkin Lymphoma (NHL); Diffuse large B-Cell lymphoma (DLBCL); Follicular lymphoma (FL); Registry; Connect®
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Collect, store, and test tumor biopsies, blood, plasma, DNA and RNA samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First relapsed/refractory diffuse large B-cell lymphoma: First relapsed/refractory diffuse large B-cell lymphoma (DLBCL) participants must have been diagnosed with relapsed/refractory (R/R) disease within 90 days prior to study enrollment and must intend to initiate 2L systemic treatment
- First relapsed/refractory follicular lymphoma: First relapsed/refractory (R/R) follicular lymphoma (FL) participants must have been diagnosed with R/R disease (grade 1 to 3B or transformed) within 90 days prior to study enrollment and must intend to initiate 2L systemic treatment

SUMMARY:
The Connect® Lymphoma Disease Registry is a US-based, multicenter, prospective observational (non-interventional) cohort study designed to collect real-world, participant-level data longitudinally in participants diagnosed with various subtypes of non-Hodgkin lymphoma (NHL).

DETAILED DESCRIPTION:
This Disease Registry is designed to capture the patient characteristics, practice patterns, and therapeutic strategies evaluated in community and academic centers when treating relapsed/refractory (R/R) diffuse large B-cell lymphoma (DLBCL), and R/R follicular lymphoma (FL). The data collected in this Registry will facilitate the evaluation of the current treatment landscape for non-Hodgkin lymphoma (NHL), including the clinical effectiveness, safety. No investigational product or drug will be administered as part of this study. Enrolled patients will receive treatment and evaluations for their disease according to the standard of care and routine clinical practice at each study site. All treatments that patients receive for their disease will be recorded, including any previous lymphoma treatments. Clinical outcomes will be documented as part of an objective clinical assessment. In addition, patient-reported health-related quality of life (HRQoL) outcomes data will be collected from patients using various validated instruments. Social support data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥18 years of age at the time of consent
* Must be able to provide written informed consent personally or by legally authorized representative
* Must have 1 of the following histologically confirmed Non-Hodgkin Lymphoma (NHL) subtypes:

  * Diffuse large B-cell lymphoma (DLBCL), NOS; or DLBCL high-grade lymphoma, not otherwise specified (NOS); or DLBCL high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements with DLBCL histology (double/triple-hit lymphoma)

    * Epstein-Barr virus-positive or composite DLBCL are allowed
  * Follicular lymphoma (FL)
* Must have been previously treated with ≥ 1 prior systemic therapy (e.g., chemotherapy, immunotherapy, or chemoimmunotherapy)
* For first relapsed/refractory (R/R) DLBCL cohort, participant must have confirmed R/R disease within 90 days prior to study enrollment and must intend to initiate 2L systemic treatment
* For first R/R FL cohort, participant must have confirmed R/R disease (grade 1 to 3B or transformed) within 90 days prior to study enrollment and must intend to initiate 2L systemic treatment
* Participant must be willing and able to complete enrollment and follow-up health-related quality of life (HRQoL) and social support instruments
* Participants volunteering for the Tissue Sub-Study must consent for use of their blood/tumor biopsies, which were collected as per standard of care, for exploratory analyses

Exclusion Criteria:

* Participant whose prior start and end date of DLBCL or FL treatment, and prior treatment received, including chemotherapy, radiation, surgery (not including excisional biopsies), and other anticancer therapy, are unknown
* Participant who has any other active malignancy (non-DLBCL or non-FL) for which the participant is receiving treatment at the time of enrollment or any other former malignancy that was diagnosed within 6 months prior to Registry enrollment (with the exception of non-melanoma skin cancer)
* Currently enrolled in any interventional clinical trial where the participant is being treated with an investigational product that cannot be identified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive participants with confirmed relapsed/refractory (R/R) diffuse large B-cell lymphoma (DLBCL) or follicular lymphoma (FL) will be screened for eligibility and enrolled from approximately 100 sites in the United States, consisting mainly of community oncology sites (~80%) and academic sites (~20%) throughout the United States. A total of approximately 1000 participants will be enrolled over an estimated 3-year period in the Registry into 1 of the 2 predefined cohorts listed above.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Patient characteristics | Up to 5 years
  Describe patient characteristics in community and academic settings
Diagnostic and Treatment Patterns - Treatment Sequencing | Up to 5 years
  Describes treatment sequencing
Progression-free Survival (PFS) | Up to 5 years
  Evaluate the effectiveness of various treatments on progression-free survival (PFS)
Event-free Survival (EFS) | Up to 5 years
  Evaluate the effectiveness of various treatments on event free survival (EFS)
Overall Response Rate (ORR) | Up to 5 years
  Evaluate the effectiveness of various treatments on the overall response rate (ORR)
Time to Next Treatment (TTNT) | Up to 5 years
  Evaluate the effectiveness of various treatments on time to next treatment (TTNT)
Overall Survival (OS) | Up to 5 years
  Evaluate the effectiveness of various treatments on Overall Survival (OS)
Practice patterns | Up to 5 years
  Describe practice patterns in community and academic settings
Therapeutic strategies | Up to 5 years
  Describe therapeutic strategies in community and academic settings
Diagnostic and Treatment Patterns - Changing Treatment Landscape | Up to 5 years
  Describes changing treatment landscape over time
Diagnostic and Treatment Patterns - Factors Associated with Treatment Choice | Up to 5 years
  Describes factors associated with treatment choice, including CAR T-cell and non-CAR T-cell therapies

SECONDARY OUTCOMES:
Safety Outcomes | Up to 5 years
  Describe safety outcomes associated with treatment regimens (adverse events of interest [AEIs]and SAEs)
Healthcare Resource Utilization (HCRU) | Up to 5 years
  Describe patient-reported HRQoL outcomes among the overall cohort population and among patient subgroups of interest (e.g.,age, risk, treatment regimen, disease subtype)
Patient Reported Outcomes | Up to 5 years
  Describe patient-reported health-related quality of life (HRQoL) outcomes among the overall cohort population and among patient subgroups of interest (e.g. age, risk, treatment regimen, disease subtype)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (53):
- United States (53):
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Local Institution - 105, Hot Springs, Arkansas
  - Rocky Mountain Cancer Centers (Boulder) - USOR, Boulder, Colorado
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - Local Institution - 169, Pensacola, Florida
  - Bond Clinic, P.A., Winter Haven, Florida
  - Local Institution - 121, Winter Haven, Florida
  - Harbin Clinic, Rome, Georgia
  - Local Institution - 112, Savannah, Georgia
  - Summit Cancer Care, PC, Savannah, Georgia
  - Local Institution - 127, Urbana, Illinois
  - Cotton O'Neil Clinical Research, Hematology and Oncology, Topeka, Kansas
  - Local Institution - 133, Topeka, Kansas
  - Local Institution - 134, Lewiston, Maine
  - Local Institution - 106, Bethesda, Maryland
  - Regional Cancer Care Associates, Bethesda, Maryland
  - Local Institution - 139, Chevy Chase, Maryland
  - Local Institution - 101, Cumberland, Maryland
  - UPMC Western Maryland Corporation, Cumberland, Maryland
  - Local Institution - 130, Hyannis, Massachusetts
  - Local Institution - 110, Saint Louis Park, Minnesota
  - Oncology Research, HealthPartners Institute, Saint Louis Park, Minnesota
  - Local Institution - 119, Joplin, Missouri
  - Local Institution - 108, Lincoln, Nebraska
  - Local Institution - 162, Reno, Nevada
  - New Jersey Cancer Care, Belleville, New Jersey
  - Astera Cancer Care East Brunswick, East Brunswick, New Jersey
  - Local Institution - 132, Florham Park, New Jersey
  - Local Institution - 140, Freehold, New Jersey
  - Local Institution - 141, Howell Township, New Jersey
  - Local Institution - 138, Little Silver, New Jersey
  - Local Institution - 128, Kinston, North Carolina
  - Local Institution - 111, Canton, Ohio
  - Tri County Hematology Oncology, Canton, Ohio
  - Local Institution - 113, North Canton, Ohio
  - Local Institution - 156, Springfield, Oregon
  - Local Institution - 149, Bethlehem, Pennsylvania
  - Local Institution - 170, Philadelphia, Pennsylvania
  - Local Institution - 171, West Reading, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - Local Institution - 117, York, Pennsylvania
  - Charleston Oncology, P.A, Charleston, South Carolina
  - Local Institution - 109, Charleston, South Carolina
  - Local Institution - 118, Knoxville, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Local Institution - 125, Fort Sam Houston, Texas
  - Local Institution - 102, Houston, Texas
  - Local Institution - 103, The Woodlands, Texas
  - Renovatio Clinical (Millennium Physicians Woodlands), The Woodlands, Texas
  - Local Institution - 115, Tacoma, Washington
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Local Institution - 122, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html